CLINICAL TRIAL: NCT06558188
Title: Combined Anabolic Therapy Study
Brief Title: Combined Anabolic Therapy
Acronym: CAT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Benjamin Leder, MD, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P002279; 1R21AR083567-01A1 (NIH)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — romosozumab; Teriparatide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Romosozumab (Active Comparator): romosozumab
  Interventions: Drug: Romosozumab
- Romosozumab and Teriparatide (Active Comparator): romosozumab and teriparatide
  Interventions: Drug: Romosozumab; Drug: Teriparatide

INTERVENTIONS:
Drug: Romosozumab — romosozumab 210 milligrams monthly
  Other Names: Evenity
Drug: Teriparatide — teriparatide 20 micrograms daily
  Other Names: Forteo
  Arms: Romosozumab and Teriparatide

SUMMARY:
In this research study the study investigators want to learn more about the effect of two different FDA-approved medication regimens in the treatment of postmenopausal osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* women aged 45+
* postmenopausal
* osteoporotic with high risk of fracture

Exclusion Criteria:

* no significant previous use of bone health modifying treatments
* known congenital or acquired bone disease other than osteoporosis
* significant renal disease, liver disease, cardiopulmonary disease, or psychiatric disease
* abnormal calcium or parathyroid hormone level
* serum vitamin D <20 ng/dL
* anemia (hematocrit <32%)
* history of malignancy (except non-melanoma skin carcinoma)
* excessive alcohol use or substance abuse
* known contraindications to romosozumab or teriparatide

Min Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 50 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Lumbar spine areal bone mineral density | Month 0 to 12
  Change in lumbar spine bone density between month 0 and month 12

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Leder, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided